CLINICAL TRIAL: NCT00016055
Title: Interleukin 12-Primed Activated T Cells As Therapy For Patients With Metastatic Melanoma (Phase I)
Brief Title: Biological Therapy and Temozolomide in Treating Patients With Metastatic Melanoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Luke's Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068590; STLMC-IMM-0002; NCI-V01-1657
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2006-11

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Temozolomide

INTERVENTIONS:
Biological: lymphokine-activated killer cells
Drug: temozolomide

SUMMARY:
RATIONALE: Biological therapies use different ways to stimulate the immune system and stop cancer cells from growing. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining biological therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of biological therapy combined with temozolomide in treating patients who have metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of interleukin-12-primed activated T cells (12ATC) and temozolomide in patients with metastatic melanoma.
* Determine the maximum tolerated dose of 12ATC in this patient population.
* Determine the clinical response of patients treated with this regimen.

OUTLINE: This is a dose-escalation study of interleukin-12-primed activated T cells (12ATC).

Patients undergo leukopheresis on days 1-3 until adequate peripheral blood mononuclear cells (PBMC) are obtained. The PBMC are treated in vitro over 2 weeks with monoclonal antibody anti-CD3, interleukin-2, and interleukin-12 to form 12ATC.

Patients receive oral temozolomide on days 15-19 and 43-47 and 12ATC IV over 15-30 minutes on days 22, 25, 29, 32, 36, 39, 50, 53, 57, 60, 64, and 67 in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of 12ATC until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 patients experience dose-limiting toxicity.

Patients are followed weekly for 2 weeks, every 3 months for 1 year, and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 9-18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic melanoma

  * No ocular or mucosal melanoma
* Must meet one of the following criteria:

  * Failed standard or salvage therapy
  * Ineligible for standard therapy due to concurrent illness
  * Declined standard therapy
* Received at least 1 prior therapy for metastatic disease
* Brain metastasis as only site of metastatic disease allowed if there is documented evidence of progression after at least 1 prior treatment for metastases
* No leptomeningeal metastases
* At least 1 documented site of bidimensionally measurable disease by MRI or CT scan

  * Previously irradiated lesions not considered measurable unless documented disease progression after radiotherapy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL
* No coagulation disorder such as thrombophlebitis

Hepatic:

* Bilirubin less than 2.0 mg/dL
* AST and ALT less than 3 times upper limit of normal (ULN)
* Alkaline phosphatase less than 3 times ULN

Renal:

* Creatinine less than 1.5 times ULN
* BUN less than 1.5 times ULN

Cardiovascular:

* Ejection fraction at least 45%
* No active ischemia
* No unstable angina
* No uncontrolled congestive heart failure

Pulmonary:

* Normal pulmonary function tests within the past month
* FEV1 or FVC more than 65% predicted
* No uncontrolled pulmonary embolism

Gastrointestinal:

* No frequent vomiting
* No medical condition that would preclude oral medication intake (e.g., partial bowel obstruction)

Other:

* No prolonged grade 4 myelosuppression from prior dacarbazine lasting more than 3 weeks
* No uncontrolled cortical dysfunction
* No other major medical illness (e.g., active systemic infection, autoimmune disease, or uncontrolled thyroid abnormality)
* No other malignancy within the past 5 years except resected basal cell carcinoma or carcinoma in situ of the cervix
* No significant psychiatric disease that would preclude study compliance
* No AIDS-related illness
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Biologic therapy:

* More than 1 month since prior biologic therapy or immunotherapy

Chemotherapy:

* More than 1 month since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)

Endocrine therapy:

* At least 4 weeks since prior steroid therapy or steroid-containing compounds
* At least 2 weeks since prior topical or inhaled steroids

Radiotherapy:

* See Disease Characteristics
* More than 1 month since prior radiotherapy, interstitial brachytherapy, or radiosurgery

Surgery:

* At least 1 week since prior surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2000-11

PRIMARY OUTCOMES:
Maximum tolerated dose at completion of study
Safety as measured by NCI common toxicity table at completion of study

CONTACTS AND LOCATIONS:
Overall Officials: John P. Hanson, MD, Study Chair — St. Luke's Medical Center
Locations (1):
- Vince Lombardi Cancer Clinic at Aurora St. Luke's Medical Center, Milwaukee, Wisconsin, United States